CLINICAL TRIAL: NCT00627276
Title: Omega-3 Fatty Acids and Prevention of DCIS and/or ADH: A Translational Approach
Brief Title: Omega-3 Fatty Acids in Treating Women With Newly Diagnosed Ductal Carcinoma In Situ and/or Atypical Ductal Hyperplasia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: OHSU Knight Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Jackie Shannon, Principal Investigator, OHSU Knight Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CDR0000581419; P30CA069533 (NIH); OHSU-3872 (Other: OHSU IRB); OHSU-CTRC-1037 (Other: OHSU OCTRI CTRC number); NCI-2013-00768 (Registry Identifier: Clinical Trials Reporting Program (CTRP))
Record Dates: First submitted 2008-02-29; First posted 2008-03-03 (Estimated); Last update posted 2017-04-27 (Actual); Status verified 2015-07

CONDITIONS: Breast Cancer; Precancerous Condition
Keywords: ductal breast carcinoma in situ; atypical ductal breast hyperplasia
MeSH Terms: conditions — Breast Neoplasms; Precancerous Conditions; Carcinoma, Intraductal, Noninfiltrating | interventions — Fatty Acids, Omega-3

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (Experimental): Patients receive oral omega-3 fatty acid capsules 3 times daily for up to 8 weeks.
  Interventions: Dietary Supplement: omega-3 fatty acid
- Arm II (Placebo Comparator): Patients receive oral placebo olive oil capsules 3 times daily for up to 8 weeks.
  Interventions: Other: placebo

INTERVENTIONS:
Dietary Supplement: omega-3 fatty acid — Oral, 3 times daily
  Arms: Arm I
Other: placebo — Oral, 3 times daily
  Arms: Arm II

SUMMARY:
RATIONALE: Polyunsaturated fatty acids are important for normal growth and development. One type, called omega-3 fatty acids (found in fish, fish oil, and some other foods), may affect the growth of abnormal breast cells.

PURPOSE: This randomized pilot trial is studying how well omega-3 fatty acids work in treating women with newly diagnosed ductal carcinoma in situ and/or atypical ductal hyperplasia.

DETAILED DESCRIPTION:
OBJECTIVES:

* To determine the effect of omega-3 fatty acids on markers of breast cancer progression in women with newly diagnosed ductal carcinoma in situ and/or atypical ductal hyperplasia.
* To determine the effect of omega-3 fatty acids on specific targets identified by microarray in breast cancer cells and in primary cultures from benign and malignant breast tissue biopsies.

OUTLINE: This is a multicenter study. Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive oral omega-3 fatty acid capsules 3 times daily for up to 8 weeks.
* Arm II: Patients receive oral placebo olive oil capsules 3 times daily for up to 8 weeks.

Patients complete questionnaires at baseline, weekly during study treatment, at the completion of study treatment, and then at 30 days after completion of study treatment. These questionnaires include the Fish Oil Adverse Event Questionnaire, the Diet and Family History Questionnaire, the Changes to Diet and Medications Questionnaire, and the Post-Intervention Questionnaire.

Patients undergo blood, urine, nipple aspirate, and tissue sample collection at baseline and after completion of study treatment for translational research studies. Blood samples are analyzed for genetic markers for breast cancer risk and progression by microarray analysis and red blood cell (RBC) fatty acids. Nipple aspirate samples are analyzed for fatty acids to determine the extent to which omega-3 fatty acid supplementation alters the fatty acid profile of breast tissue. Tissue samples are analyzed for the presence of ductal carcinoma in situ and/or atypical ductal hyperplasia or invasive cancer. Leftover blood, urine, nipple aspirate, and tissue samples are stored for future research studies.

After completion of study treatment, patients are followed at 30 days.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Biopsy confirmed diagnosis of any of the following:

  * Ductal carcinoma in situ (DCIS) and/or atypical ductal hyperplasia (ADH)
  * DCIS with a component of invasive carcinoma
  * ADH with a component of invasive carcinoma
  * DCIS and ADH with a component of invasive carcinoma
* Newly diagnosed disease
* No pure invasive breast cancer on biopsy without a component of DCIS or ADH
* Hormone receptor status not specified

PATIENT CHARACTERISTICS:

* Female
* Menopausal status not specified
* Not pregnant
* Negative pregnancy test
* Speaks English or Spanish
* No allergy to fish oil or olive oil
* No condition that, in the opinion of the study clinician, would make participation in the study harmful to the patient

PRIOR CONCURRENT THERAPY:

* No concurrent therapeutic anticoagulation
* No concurrent use of fish oil > 1 g/day

Ages: 21 Years to 120 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2007-12; Primary Completion 2012-12 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Effect of omega-3 fatty acids on markers of breast cancer progression | minimum 2 weeks, maximum 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jackilen Shannon, PhD, Principal Investigator — OHSU Knight Cancer Institute
Locations (2):
- United States (2):
  - Epic Imaging, Portland, Oregon
  - Knight Cancer Institute at Oregon Health and Science University, Portland, Oregon